CLINICAL TRIAL: NCT02464501
Title: The COPPER-A Trial: The Occlusion Perfusion Catheter for Optimal Delivery of Paclitaxel for the Prevention of Endovascular Restenosis - Above and Below the Knee
Brief Title: The OPC for Optimal Delivery of Paclitaxel for the Prevention of Endovascular Restenosis - Above and Below the Knee
Acronym: COPPER-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horizons International Peripheral Group (Other)
Collaborators: Advanced Catheter Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIPG-CLIN-2015-02
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Peripheral Arterial Disease; Cardiovascular Disease; Peripheral Vascular Disease
Keywords: PAD; COPPER-A; Peripheral Arterial Disease; OPC; Occlusion Perfusion Catheter; Paclitaxel; Pressana; Precision Delivery System
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- OPC Treatment (Experimental): Paclitaxel administration using the OPC for the prevention of restenosis in infrainguinal de novo and restenotic femoropopliteal lesions. Subjects will be treated with the endovascular intervention selected by the treating physician in reference vessels ranging from 4mm to 7mm in diameter. Following the achievement of optimal interventional results (less than thirty (30) percent residual stenosis without stenting) the OPC will be placed at the interventional treatment area and paclitaxel will be delivered to the treated segment. Data will be collected to assess acute safety, long-term safety and durability to demonstrate the safety and efficacy of paclitaxel delivered with the ACT, Inc. OPC device.
  Interventions: Other: Paclitaxel administration using the OPC

INTERVENTIONS:
Other: Paclitaxel administration using the OPC

SUMMARY:
The purpose of this study is to assess the safety and efficacy of paclitaxel administration using the occlusion perfusion catheter (OPC) for the prevention of restenosis in infrainguinal de novo, restenotic femoropopliteal and infrapopliteal stenoses and occlusions, and in-stent restenosis.

DETAILED DESCRIPTION:
The purpose of this study is to assess the safety and efficacy of paclitaxel administration using the occlusion perfusion catheter (OPC) for the prevention of restenosis in infrainguinal de novo, restenotic femoropopliteal and infrapopliteal stenoses and occlusions, and in-stent restenosis. Subjects will be treated with the endovascular intervention selected by the treating physician in SFA reference vessels ranging from 4mm to 7mm in diameter and infrapopliteal vessels ranging from 2mm to 4mm. Following the achievement of optimal interventional results (less than thirty (30) percent residual stenosis without stenting) the OPC will be placed at the interventional treatment area and paclitaxel will be delivered to the treated segment. Data will be collected to assess acute safety, long-term safety and durability to demonstrate the safety and efficacy of paclitaxel delivered with the ACT, Inc. OPC device.

ELIGIBILITY:
General Inclusion Criteria:

* Willing and able to provide informed consent and comply with all study requirements;
* Candidate for peripheral vascular femoropopliteal or infrapopliteal percutaneous intervention;
* Must be ≥ 18 years of age;
* Rutherford category 2, 3, 4, or 5;
* Willing and able to tolerate dual anti-platelet therapy (DAPT) for a minimum of one (1) month;
* Lab work within acceptable limits according to standard of care;
* INR < 2.0 if on warfarin or not on warfarin;
* Minimum sheath size used for the interventional procedure

  * 7x8 OPC Catheter - 7FR.
  * 3x15 OPC, 3x15 PRESSANA(TM), or 3x8 PRESSANA(TM) - 6FR.

General Exclusion Criteria:

* Life expectancy < three (3) years;
* Planned amputation prior to procedure;
* Pregnancy or nursing (a pregnancy test is required for all women of childbearing capabilities ≤ 7 days prior to the index procedure);
* Previous intervention of the target lesion with a drug eluting balloon or drug delivery catheter;
* Any treatment in the target vessel with drug eluting balloon;
* Acute limb ischemia
* Known allergy to paclitaxel;
* Known hypersensitivity to other drugs manufactured in Cremophor® EL (polyoxyethylated castor oil; e.g. Drugs containing polyoxyethylated castor oil are drugs such as miconazole, cyclosporine injection, nelfinavir mesylate, saperconazole, tacrolimus, and xenaderm ointment);
* Known allergy to anticoagulants;
* Known TRUE acetylsalicylic acid (ASA) allergy;
* Use of glycoprotein (GP) IIb/IIIa inhibitors during the procedure visit within 30 days following the index procedure;
* Target lesion treated with a cryoplasty balloon at the time of the index procedure;
* Hemorrhagic stroke within six (6) months;
* Renal failure or chronic kidney disease with GFR ≤30 mL/min or MDRD GFR ≤30 mL/min per 1.73 m2 (or serum creatinine ≥2.5 mg/L within 30 days of index procedure or treated with dialysis);
* Prior vascular surgery of the index limb;
* Current enrollment in another investigational device or drug study;
* After obtaining informed consent, at any point up to introduction of the OPC, the investigator determines the study subject is not appropriate for the study.

Angiographic Inclusion Criteria:

* Reference vessel diameter (RVD) ≥ 4 mm and ≤ 7 mm for femoropopliteal arteries or ≥ 2 mm and ≤ 4 mm for infrapopliteal arteries;
* Either single or multiple lesions in the SFA and/or popliteal artery or single or multiple lesions in the infrapopliteal arteries (AT, PT, peroneal);
* For single lesion treatment, minimum lesion length ≥ 20 mm;
* Minimum of one patent infrapopliteal vessel;
* Pre-intervention percent DS ≥ 70%.

Angiographic Exclusion Criteria:

* Flow limiting dissection necessitating stent placement prior to OPC use;
* Post PTA residual stenosis ≥ 30% as visualized by treating physician;
* Perforation requiring a covered stent;
* For femoropopliteal target lesion or occlusion location extends distally beyond the P2 region of the popliteal artery or infrapopliteal lesion or occlusion location is at or proximal to the origin of the trifurcation vessel or below the ankle (top of the talus bone);
* Target lesion within a fractured stent;
* Target lesion within a stent and restenosed two (2) or more times;
* Significant (≥ 50% DS) inflow lesion or occlusion left untreated in the ipsilateral Iliac, SFA, or popliteal artery proximal to the target lesion;
* A lesion treated distal to the target lesion results in compromising inline flow distal to the target lesion;
* Visible thrombus in the target artery or proximal to the target artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Primary Patency | 12 months
  Femoropopliteal Lesions: Measured by duplex Doppler ultrasound (DUS) - demonstrated by Peak Systolic Velocity Ratio (PSVR) ≤ 2.5 and clinically free from Target Lesion Revascularization.
Primary Patency | 6 months
  Infrapopliteal Lesions: Measured by duplex Doppler ultrasound (DUS) - demonstrated by freedom from target lesion occlusion and clinically free from Target Lesion Revascularization.
Freedom from major adverse events (MAEs) | 1 month
  MAEs are defined as target limb related death, major amputation in the target limb (amputation above the metatarsals), or target lesion revascularization (TLR) within one (1) month.

SECONDARY OUTCOMES:
Primary Patency | 6 months
  Femoropopliteal Lesions: Measured by duplex Doppler ultrasound (DUS) - demonstrated by Peak Systolic Velocity Ratio (PSVR) ≤ 2.5 and clinically free from Target Lesion Revascularization.
Primary Patency | 12 months
  Infrapopliteal Lesions: Measured by duplex Doppler ultrasound (DUS) - demonstrated by freedom from target lesion occlusion and clinically free from Target Lesion Revascularization.
Improvement in Rutherford category | 3, 6, and 12 months
Primary Assisted Patency | 1, 3, 6, and 12 months
  Patency of the target lesion following endovascular re-intervention of the target lesion due to symptomatic restenosis.
Secondary Patency | 1, 3, 6, and 12 months
  Measured by patency of the target lesion after treatment of a (re)occlusion of the index lesion during the follow-up period.
Freedom from target lesion revascularization (TLR) | 1, 3, 6, and 12 months
Freedom from target vessel revascularization (TVR) | 1, 3, 6, and 12 months
Improvement in Walking Impairment Questionnaire scores | 6 and 12 months
Device Success | Day 1 - Index Procedure
  Defined as the ability to deliver paclitaxel to the interventional treatment length as intended.
Freedom from major adverse events (MAEs) | 1, 3, 6, and 12 months
Anticipated adverse events | 1, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank Bunch, MD, FACC, Principal Investigator — Cardiology Associates
Locations (17):
- United States (17):
  - Cardiology Associates, Fairhope, Alabama
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - Vascular Institute of the Midwest, Davenport, Iowa
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Michigan Outpatient Vascular Institute, Dearborn, Michigan
  - St. John Hospital, Detroit, Michigan
  - Mid-Michigan Heart & Vascular Center, Saginaw, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Novant Health, Charlotte, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - University Surgical Associates, Chattanooga, Tennessee
  - Kore Cardiovascular Research, Jackson, Tennessee
  - Huntsville Memorial Hospital, Huntsville, Texas
  - North Dallas Research Associates, McKinney, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No